CLINICAL TRIAL: NCT04549350
Title: Sleep Quality Among Health Care Workers During COVID-19 Pandemic: Kuwait Experience
Brief Title: Sleep Quality Among HCWs
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Collaborators: Ministry of Health, Kuwait (Other Government)
Responsible Party: Principal Investigator, Ahmad Abbas, Lecturer of chest diseases, Zagazig University
Other Study IDs: 2020/1464
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PSQI — Assessment of sleep quality using Pittsburgh Sleep Quality Index (PSQI): It is a simple tool which assess the sleep quality over one month period. It included seven components with a global PSQI score > 5 is indicative of poor sleep quality

SUMMARY:
The novel coronavirus has brought the world into uncharted waters. Whole countries are on lockdown, the economy has ground to a halt, and many people are afraid for themselves and their loved ones. With such unprecedented changes coming on so quickly, it's understandable that the importance of sleep is flying under the radar. But as we adjust to stay-at-home orders and try to remain healthy in a time of COVID-19, focusing on sleeping well offers tremendous benefits.

Millions of people suffered from insomnia before the coronavirus, and unfortunately, the pandemic creates a host of new challenges even for people who previously had no sleeping problems. The coronavirus pandemic doesn't affect everyone in the same way. Of course, patients with the virus and front-line medical workers face the brunt of the direct impacts of the disease. Social distancing, school closures, quarantines, working-from-home: all bring profound changes to normal routines for people of all ages and walks of life.

The aim of the current work is to assess the sleep quality among health care workers in the front-line management of COVID-19 in Kuwaiti Ministry of Health hospitals and its relation on medical errors.

ELIGIBILITY:
Inclusion Criteria:

-Health care workers at Kuwait Ministry of Health hospitals during the period from May 2020 to July 2020

Exclusion Criteria:

* Care givers above 60 years
* those who refuse to participate or requested to withdraw from the study at any time
* HCWs who were not on duty at the time of survey due to any leave or absence
* replies with incomplete answers or duplicate answers

Ages: 25 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Health care workers (HCWs) at Kuwaiti Ministry of Health hospitals ,Kuwait during the period from May 2020 to July 2020
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-09-05 (Actual)

PRIMARY OUTCOMES:
Presence of poor sleep quality or not | one month period
  survey

SECONDARY OUTCOMES:
reported medical errors | one month
  survey

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, Egypt